CLINICAL TRIAL: NCT03563404
Title: Are Portal Blood Flushes Useful in Maintaining Hemodynamic Stability in the Peri-Reperfusion Stage of Orthotopic Liver Transplantation
Brief Title: Portal Blood Flushes in the Peri-Reperfusion Stage of Liver Transplantation
Status: Completed | Type: Observational
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00044952
Record Dates: First submitted 2016-05-03; First posted 2018-06-20 (Actual); Last update posted 2018-07-03 (Actual); Status verified 2018-07

CONDITIONS: Liver Disease
MeSH Terms: conditions — Liver Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Portal Blood Flush: participants that receive the portal blood flush
- No Portal Blood Flush: participants that don't receive the portal blood flush

SUMMARY:
By showing that increased levels of acidotic metabolites and electrolytes in the systemic blood of patients who do not receive portal blood flush prior to reperfusion compared to patients who do receive portal blood flush, and that these increased levels correlate with cardiac depression as seen on TEE, the investigators hope to find a superior technique for liver reperfusion.

ELIGIBILITY:
Inclusion Criteria:

* Liver Transplantation
* 18 years old or older

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Liver Transplant
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2015-06-29; Primary Completion 2016-06-29 (Actual); Study Completion 2016-06-29 (Actual)

PRIMARY OUTCOMES:
Hemodynamic Stability | 5 days
  The primary objective of this study is to determine whether or not a portal blood flush is useful for maintaining hemodynamic stability in the peri-reperfusion stage of Orthotopic Liver Transplantation as evidence by TEE.

SECONDARY OUTCOMES:
correlation between the cardiac dysfunction and the degree of hyperkalemia seen after reperfusion. | 5 days
  The secondary objective is to determine if there is a correlation between cardiac dysfunction as measured by a qualitative analysis of TEE and the degree of hyperkalemia measured by a post reperfusion blood sample.

CONTACTS AND LOCATIONS:
Overall Officials: Grayce Davis, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States